CLINICAL TRIAL: NCT03119077
Title: Randomized, Double-blind, Placebo-controlled, Escalating Single Dose Study of the Safety, Tolerability, and Pharmacokinetics of Orally Administered BAY1161116 in Healthy Postmenopausal Women Including Food-effect and Drug-drug-interaction With Itraconazole
Brief Title: Single Ascending Dose, First-in-Human Study on Safety, Tolerability and Pharmacokinetics of BAY1161116
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study early terminated due to lower drug exposure
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 18752; 2016-003520-23 (EudraCT Number)
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY1161116 (Experimental): Dose steps 1 to 6 of BAY1161116 (increasing dose levels)
  Interventions: Drug: BAY1161116; Drug: Itraconazole
- Placebo (Placebo Comparator): Placebo Dose 1 to 6 of BAY 1161116
  Interventions: Drug: Placebo; Drug: Itraconazole

INTERVENTIONS:
Drug: BAY1161116 — Escalating doses of BAY1161116; single dose administration; redosing of BAY1161116 at dose group 1 together with itraconazole; redosing of BAY1161116 at dose group 2 as liquid service formulation, redosing of BAY1161116 at dose group 3 together with food
  Arms: BAY1161116
Drug: Placebo — Escalating doses of respective placebos; single dose administration; redosing of placebo at dose group 1 together with itraconazole; redosing of placebo at dose group 2 as liquid service formulation, redosing of placebo at dose group 3 together with food
  Arms: Placebo
Drug: Itraconazole — Redosing of BAY1161116/placebo at dose group 1 together with itraconazole

SUMMARY:
This study will be conducted in a single center, double-blind with 6 dose escalation groups to evaluate the safety, tolerability, and pharmacokinetics of single ascending doses of BAY1161116.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female postmenopausal subjects
* Age: 45 to 65 years (inclusive)
* Body mass index (BMI) : ≥18 and ≤30 kg/m²
* Non-smoker for 3 months (former smokers who quit smoking >3 months before the first study drug administration may be included)

Exclusion Criteria:

* Incomplete recovery from pre-existing disease for which it can be assumed that the absorption, distribution, excretion,and effect of the study drugs will not be normal
* Any use of systemic or topically active medication or herbal remedies, prescription or non-prescription, from screening to the first drug administration (occasional use of paracetamol or ibuprofen is permissible)
* Any severe disease within the last 4 weeks prior to the first study drug administration
* History of orthostatic hypotension, fainting spells, blackouts
* Any malignant tumor and history thereof
* Any other medical condition which, at the discretion of the investigator, would make study participation unadvisable
* Any clinically relevant finding at the physical- and gynecological examinations
* Allergy, hypersensitivity, or non-allergic drug reactions to any excipient of the IMP or reference/interaction product
* Regular alcohol consumption equivalent to >20 g alcohol per day
* Urine screen positive for any drug or cotinine

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of TEAEs | 5 weeks
  TEAEs: treatment-emergent adverse events
Severity of TEAEs | 5 weeks
  TEAEs: treatment-emergent adverse events
AUC of BAY1161116 | 5 weeks
  AUC: Area under the concentration vs. time curve from zero to infinity
Cmax of BAY1161116 | 5 weeks
  Cmax: maximum observed drug concentration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany